CLINICAL TRIAL: NCT02871388
Title: Addressing Modifiable Breast Cancer Risk Factors With Project CONECT [Connect Online to Engage Change Tool]
Brief Title: Addressing Modifiable Breast Cancer Risk Factors With Project CONECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCC-16-12892; HM20008111 (Other: IRB)
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Weight Loss; Breast Cancer Risk Factors
Keywords: Physical activity; Diet; Nutrition; Breast cancer prevention; Mammography screening
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONECT (Experimental): 12 week program with additional follow up at 24 weeks.
  Interventions: Behavioral: CONECT
- Control (No Intervention): Waitlist control. No intervention for first 12 weeks. Participants given the option to participate in the program after 24 weeks.

INTERVENTIONS:
Behavioral: CONECT — 1 monthly in person + 1 monthly telephone + 4 monthly email contact for behavior modification. Focus on motivation, self efficacy and information provision.
  Arms: CONECT

SUMMARY:
The objective of this protocol is to adapt and pilot test an existing lifestyle modification intervention for weight loss for women with overweight or obesity who have had a recent false positive mammography screen. The purpose of this pilot trial is to establish feasibility of Connect Online to Engage Change Tool (CONECT) to promote weight loss through increased physical activity and diet change.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 40-65 years of age,
3. Received a negative mammography screening result in the previous four weeks
4. Moderately sedentary lifestyle (less than 120 minutes/week moderate intensity activity),
5. Answer "no" to all questions on the Physical Activity Readiness Questionnaire (PAR-Q).
6. BMI 25-40 kg/m2
7. Has access to a computer or mobile device with wireless internet
8. Able to speak and read English (language requirements are necessary because we cannot accommodate additional languages in prototype development phase.)

Exclusion Criteria:

1. Previous history or current diagnosis of breast cancer
2. Pregnancy or lactation
3. Involvement in a weight loss program
4. Major co-morbidities (e.g.,diabetes, hypertension, etc.)
5. History of disordered eating
6. Currently taking medication that may impact weight (e.g., synthroid, metformin)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
feasibility-participant engagement and retention | 12 weeks
  recruitment of 30 participants with 70% retention at 12 weeks
feasibility-intervention adherence | 12 weeks
  Completion of 80% of intention components including wearing Fitbit tracker, completed of the weekly weightings, answering emails, attending intervention sessions

SECONDARY OUTCOMES:
Change in autonomous motivation | 12 weeks and 24 weeks
  Motivation assessment and feedback.
Steps per day | 12 and 24 weeks
  participants will be asked to use the Fitbit Heart Rate (HR) Physical Activity Monitor to track daily steps and minutes of physical activity.
Total minutes of weekly physical activity | 12 and 24 weeks
  assessed by 7 day Physical Activity Recall Scale (PAR)
Daily caloric goals | 12 and 24 weeks
  assessed by Automated Self-Administered (ASA) 24

OTHER OUTCOMES:
change in waist circumference | 12 and 24 weeks
  waist circumference measured at 12 and 24 weeks.
weight loss | 12 weeks
  percent weight loss at 12 weeks
weight maintenance | 24 weeks
  for intervention group only, percent weight loss at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria D Thomson, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States